CLINICAL TRIAL: NCT01531049
Title: Smoking Cessation in Young Adults in Northern Finland
Brief Title: Smoking Habits and Smoking Cessation in Young Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tuula Toljamo (Other)
Collaborators: University of Oulu (Other); University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Tuula Toljamo, Chief Chest Physician, Lapland Central Hospital,Rovaniemi,Finland, University of Oulu
Organization: University of Oulu (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EETTMK:99/2011
Record Dates: First submitted 2012-02-03; First posted 2012-02-10 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Smoking Cessation; Smoking; Habits
Keywords: smoking cessation; young adults; motivational counselling; smoking; nicotine replacement therapy; therapy
MeSH Terms: conditions — Smoking Cessation; Smoking; Habits | interventions — Varenicline; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Varenicline (Experimental): A varenicline treatment group (with motivational interview technique combined with varenicline and placebo transdermal patch). Intervention with Nicorette 15mg /16 h patch
  Interventions: Drug: varenicline
- Nicotine cutaneous patch 15mg (Experimental): Intervention with Varenicline for 12 weeks. Nicotine cutaneous patch 15mg/16h
  Interventions: Drug: Nicotine cutaneous patch 15mg/16h
- Nicotine cutaneous patch 10mg (Experimental): Intervention with Placebo transdermal patch for 8 weeks. Nicotine cutaneous patch 10mg/16h
  Interventions: Drug: Nicotine cutaneous patch 10mg/16h; Other: Placebo cutaneous patch
- Placebo cutaneous patch (Placebo Comparator): No active medication.One transdermal patch/16 h.Total duration was 8 weeks.
  Interventions: Drug: Nicotine cutaneous patch 10mg/16h; Other: Placebo cutaneous patch

INTERVENTIONS:
Drug: varenicline — days 1.-3 0,5mgx1/day, days 4.-7 0,5mgx2/day, day 8 to the 12weeks 1mgx2 /day
  Other Names: Champix
  Arms: Varenicline
Drug: Nicotine cutaneous patch 15mg/16h — One patch for 16hours/day and duration of 8 weeks.
  Other Names: Nicorette
  Arms: Nicotine cutaneous patch 15mg
Drug: Nicotine cutaneous patch 10mg/16h — One patch 16hours/day and duration of 8 weeks
  Other Names: Nicorette
  Arms: Nicotine cutaneous patch 10mg; Placebo cutaneous patch
Other: Placebo cutaneous patch — No active medication.O ne patch 16hours and duration for 8 weeks
  Other Names: Leukomed T
  Arms: Nicotine cutaneous patch 10mg; Placebo cutaneous patch

SUMMARY:
The purpose of this study is to assess the efficacy and effectiveness of varenicline and nicotine patch combined with motivational interview technique in smoking cessation of young adults over 12 months follow-up.

DETAILED DESCRIPTION:
Most teenage smokers are still smoking when they become adults confirming that stopping of smoking at young age is difficult although majority of young smokers want to quit. Young smokers experience many relapses partly due to the lack of appropriate and available cessation services. The discomfort experienced during cessation attempts is likely to be negatively associated with cessation success. Quitting of smoking is by the far most important procedure in preventing COPD progression. In Finland, 18-35% of young adults smoke, the variability being associated at least with socioeconomic background, education and geographical area. Our recent studies on male military draftees have shown that smoking is much more frequent in Northern than Southern Finland. However young men want to quit and accept new smoking restrictions. Very few studies are available on quitting attempts or counselling, pharmacotherapy and/or their combinations in young adults who want to quit.

ELIGIBILITY:
Inclusion Criteria:

* healthy daily smokers
* a daily smoker has smoked at least 1cig/day every day during last month and has smoked at least 100 cig ever
* a nonsmoker has smoked less than 50 cig ever,and has not smoked at all during last month
* motivated to quit smoking and ready to 12 months follow-up
* minor allergy or mild asthma without regular medication is allowed

Exclusion Criteria:

* any chronic disease with daily medication
* known allergy to study medications(varenicline, nicotine patch,nicotine gum)
* any substance and/or alcohol abuse
* drop-outs are counted as current smokers

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12-31 (Actual); Study Completion 2016-09-02 (Actual)

PRIMARY OUTCOMES:
The abstinence rate | 3 months follow-up

SECONDARY OUTCOMES:
The saliva cotinine verified abstinence rate | 3 months follow-up
The abstinence rate | 1, 6 and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pentti Nieminen, PhD, Principal Investigator — Medical Informatics and Statistics Research Group, University of Oulu
Locations (1):
- Lapland Central Hospital, Lapland Hospital District, Rovaniemi, Finland